CLINICAL TRIAL: NCT03435757
Title: Surgical Outcomes of Decortication With or Without Calcium Phosphosilicate Putty Following Regenerative Therapy of Non-Contained Intrabony Periodontal Defects: A Randomized Controlled Clinical Study
Brief Title: Decortication With Calcium Phosphosilicate Putty in the Treatment of Non-contained Intrabony Periodontal Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: shivaliperio
Record Dates: First submitted 2018-01-30; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-01

CONDITIONS: Periodontal Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group OFD+IMP+CPS (Experimental): OFD+IMP+CPS; open flap debridement (OFD) and intramarrow penetration (IMP) plus calcium phosphosilicate putty (CPS)
  Interventions: Procedure: OFD+IMP+CPS
- Control group (OFD+IMP) (Active Comparator): OFD+IMP;open flap debridement (OFD) and intramarrow penetration (IMP)
  Interventions: Procedure: OFD+IMP

INTERVENTIONS:
Procedure: OFD+IMP+CPS — open flap debridement (OFD) and intramarrow penetration (IMP) plus calcium phosphosilicate putty
  Arms: Test Group OFD+IMP+CPS
Procedure: OFD+IMP — open flap debridement (OFD) and intramarrow penetration (IMP)
  Arms: Control group (OFD+IMP)

SUMMARY:
To overcome the disadvantage of complex morphology and availability of less favorable support to retention of graft and clot stabilization in 1-, 1-2-wall periodontal defects, it was hypothesized that placement of CPS putty having the property of being easily moldable and shaped along with decortication would provide better healing outcome as compared to decortication alone in 1-, 1-2-wall periodontal defects.

Therefore with this rationale, the present study is carried out to evaluate the treatment outcomes of decortication with and without use of CPS putty in 1- wall, 1-2-wall periodontal defects.

DETAILED DESCRIPTION:
The definite goal of periodontal regenerative therapy is to restore the tooth supporting tissues, lost as a result of inflammatory periodontal diseases and infections. Numerous treatment modalities have been described and tested, including use of non resorbable and resorbable membranes (GTR) ; autogenous bone grafts, bone allografts, xenografts and synthetic materials, and bioactive molecules (EMD) and growth factors. Furthermore researches on cell therapy and gene therapy utilization to boost the reparative potential of the wound tissues are also being carried out. Each of the treatment modalities have their own limitations and advantages.

Autogenous bone grafts having good osteogenic and osteoconductive capacity than other grafts are considered to be the best but need for a second surgery, postoperative complaints and insufficient amount of bone graft obtained restrict their use. Allografts and xenografts use is also limited because of their controversial osteoinduction capability, ethical problems, infections and immunological rejection risk. As a result of the varying disadvantages of the auto-, allo- and xenografts, synthetic bone graft use is slowly increasing. These have advantages of good osteoconductivity, no ethical or problems of infection and production of these grafts can be unlimited. The disadvantages lies in their lack of osteogenic and osteoinductive properties.

One such synthetic material is bioactive glass developed by Hench and West In late 1960s. It is available in particulate as well as putty form. Calciumphosphosilicate (CPS) putty (NOVABONE Dental Putty, Novabone products Pvt. Ltd., INDIA) is a new next generation bone graft material built with bioactive glass platform with additives like polyethylene glycol and glycerin to improve handling and efficiency. It is available as a premixed pliable cohesive material. It's not only an osteoconductive material but also imparts osteostimulative effect. CPS putty stimulates osteoblast recruitment, proliferation and differentiation at the defect site and increases rate of bone formation throughout the defect, simultaneously increasing the resorption rate of the graft material. Bembi et al. reported that mean percentage change in amount of radiographic bone fill was more in the treatment of intrabony defects with novabone putty as compared to calcified algae- derived porous hydroxyapatite bone graft. In another study Biswas et al. concluded that use of bioactive glass osteostimulative biomaterial yields superior clinical results, including increased pocket depth reduction of class II furcation defects as compared to an autologous platelet concentrate.

Controversial reports have been reported on outcomes of healing in reference to number of bony walls remaining. Therefore type of periodontal defect might influence the effect of grafts and membrane on periodontal regeneration. Contained intrabony periodontal defects (3- walled) offer a higher predictability in the regenerative procedures as compared to non-contained infrabony periodontal defects (1-,2- wall defects) as the later morphology is complex due to limited buccal and lingual periodontal tissue component. The one wall periodontal defect offers less favorable support to the flap and clot stabilization,. Studies have shown considerable variations of results as these defects have larger width (as compared to 3-wall defects); osteoconductivity is difficult to obtain; blood supply to the gingival flap at the graft site is insufficient and gingival recession tends to occur. Selvig et al. reported that the percentage of 3-wall intrabony defect was less than 30% and a combination of 1-wall and 2- wall defects was mainly observed. The prevalence of later is more hence development of predictable periodontal regeneration holds a greater importance in these cases.

MATERIALS AND METHODS

STUDY DESIGN

This randomized controlled study will be conducted in Department of Periodontics and Oral Implantology, Post Graduate Institute of Dental Sciences, Rohtak.

STUDY POPULATION

Patients will be recruited from regular outpatient department of the Department of Periodontics and Oral Implantology and Department of Oral medicine, Diagnosis and Radiology.

The study population will consist of a minimum of 36 systemically healthy patients aged 28 to 60 years with chronic periodontitis and having at least one tooth with non-contained periodontal osseous defect (1-wall, 2-wall defect). In each patient, one non-contained bone defect will be selected, in case of more than one defect, the defect which is at the deepest in the radiographic and clinical examination will be selected, without stratification by tooth type or location. Patients will be randomized into two groups (minimum 18 each) into test and control group. Control group will undergo treatment with open flap debridement (OFD) and intramarrow penetration (IMP) (OFD+IMP; control group) and test group OFD plus IMP plus calcium phosphosilicate putty (CPS) (OFD+IMP+CPS; test group). Prior written informed consent will be taken from all the participants after explaining the study objectives and procedures in patient's own language.

METHODOLOGY

The study will be conducted as follows:

Presurgical therapy: which will include:

i. Oral hygiene instructions

ii. Full mouth supragingival and subgingival scaling and root planning with ultrasonic scaler, hand scaler and curettes.

Subjects will be re-evaluated and those satisfying the inclusion criteria will be recruited

CLINICAL PARAMETERS

Assessed Using UNC 15 periodontal probe to measure PPD, CAL, BOP, REC at 6 sites (mesial, distal, median points at buccal and lingual aspects) per tooth and at 4 sites per tooth to measure PI, GI.

1. Full mouth indices to be recorded at baseline

   Bleeding on probing (BOP)

   Probing Pocket depth (PPD)

   Clinical Attachment loss (CAL)
2. Site specific indices (6 sites per tooth)

Plaque index (PI)

Gingival index (GI)

Probing Pocket depth (PPD) - measured from gingival margin to the base of pocket

Clinical attachment loss (CAL) - measured from cementoenamel junction(CEJ) to base of the pocket

Keratinized tissue width (KTW) - distance from gingival margin to mucogingival junction (MGJ)

Gingival recession (REC) - distance in millimetres from the gingival margin to CEJ

Bleeding on probing (BOP)

Tooth mobility

RADIOGRAPHIC PARAMETERS:

Customized bite blocks and long cone paralleling technique will be used to obtain standardized radiographs.

Radiographic defect depth (rDD) - the distance from the projection on the root surface of the most coronal point of the residual bone crest to the bottom of the defect.

Radiographic defect width (rDW) - the distance from the most coronal point of the residual bone crest to the root surface, were measured using a caliper and recorded to the nearest mm.

Radiographic defect angle (ANG) - line tangential to the root surface and a line connecting the bottom of the defect to the most coronal part of the crest next to the adjacent tooth.

All radiographic parameters will be analyzed at baseline, at 6 months and at 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic periodontitis
* Presence of non- contained osseous defect
* Age 28 to 60 years (both males and females)
* Completed etiological periodontal therapy (oral hygiene instructions and scaling and root planing under local anaesthesia.
* At re-evaluation full mouth plaque score67 < 1, full mouth bleeding score FMBS <20%
* Non-smokers (Current and past smokers)
* Presence of ≥ 2mm of keratinized tissue to allow flap management

Tooth defect criteria:

* Probing pocket depth ≥ 5mm
* Clinical attachment loss ≥ 5mm
* Associated with a 1-wall, 2-wall or a combined 1-2 wall osseous defect ≥ 3mm deep located in the interproximal area of single- and multirooted teeth (assessed by transgingival probing and radiograph, further to be confirmed after flap elevation)
* Tooth mobility ≤ 1
* Concerned tooth and adjoining teeth to be vital and without symptoms or signs of endodontic involvement
* Tooth and adjoining teeth free of caries or inadequate restorations/ unrestorable tooth.
* Absence of non-working interferences.
* Interproximal intrabony defects not extending into the furcation area of molar teeth.

Exclusion Criteria:

* Medical conditions interfering with periodontal health or wound healing
* Systemic illness known to affect the periodontium or outcome of periodontal therapy.
* Patient taking medications such as corticosteroids or calcium channel blockers, which are known to interfere periodontal wound healing or patient on long term NSAID therapy.
* Patients allergic to medication (local anaesthetic, antibiotics, NSAID).
* Pregnant or lactating women.
* Fractured/perforated roots.
* Developing permanent tooth.
* History of recent periodontal treatment within 6 months prior to study.
* 3-wall intrabony defects

Ages: 28 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Bone fill, | 12 months
  bone growth fill in mm
CAL | 12 months
  clinical attachment level gain in mm

CONTACTS AND LOCATIONS:
Overall Officials: SHIVALI SAHARAN, Principal Investigator — Post Graduate Institute of Dental ISciences, rohtak
Locations (1):
- Shikha Tewari, Rohtak, Haryana, India